CLINICAL TRIAL: NCT05934838
Title: A Feasibility Trial of Tazemetostat Plus CAR T Cell Therapy in B-cell Lymphomas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Epizyme, Inc. (Industry); Applebaum Foundation (Unknown); American Society of Clinical Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-07025095
Record Dates: First submitted 2023-06-28; First posted 2023-07-07 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Follicular Lymphoma; B-Cell Lymphoma; Mantle Cell Lymphoma; Diffuse Large B Cell Lymphoma
Keywords: CAR T-cell; Tazemetostat; FL; MCL; DLBCL
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, B-Cell; Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse | interventions — tazemetostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tazemetostat and CAR T-Cell Therapy (Experimental): Tazemetostat is being administered prior to, and following, standard of care CAR T cell therapy. The use of tazemetostat in this way is investigational.
  Interventions: Drug: Tazemetostat Pill

INTERVENTIONS:
Drug: Tazemetostat Pill — Participants will take 800 mg of tazemetostat twice a day starting 7 days before apheresis and continue to take tazemetostat until lymphodepletion, which is chemotherapy given prior to receiving the CAR T cells. Participants will stop taking tazemetostat after lymphodepletion until after CAR T cell infusion. Once lymphocyte counts increase, tazemetostat will be resumed and tazemetostat will be taken for 6 - 12 months, depending on participant response.
  Other Names: Tazverik

SUMMARY:
This is a clinical trial to evaluate the feasibility and safety of giving tazemetostat followed by standard of care CAR T cell infusion in previously treated diffuse large b-cell lymphoma (DLBCL), follicular lymphoma (FL), and mantle cell lymphoma (MCL). The investigators hypothesis is that this combination has the potential to significantly improve the ability of CART cells to recognize and kill lymphoma cells without a significant impact on safety. Participants will receive the tazemetostat pills before and after receiving their CAR T cell therapy, for up to 12 months after CAR T cell administration. Patients will be followed for up to 5 years.

DETAILED DESCRIPTION:
This is a single arm, open label, clinical trial to evaluate the feasibility and safety of oral tazemetostat followed by standard of care CAR T cell infusion in previously treated DLBCL, FL, and MCL. The investigators hypothesis is that this combination has the potential to significantly improve the ability of CART cells to recognize and kill lymphoma cells without a significant impact on safety.

Tazemetostat 800 mg will be given twice daily by mouth for at least 1 week prior to apheresis, during the period between apheresis and CAR T infusion, and following lymphodepletion chemotherapy until Day 7 post-CAR T therapy. Once patients' platelets and neutrophil counts recover, tazemetostat will be resumed. Tazemetostat treatment will continue for up to 6 months in patients with complete responses and up to 12 months in patients with partial responses.

A 3+3 trial design will be implemented for the first six patients enrolled. The regimen will be considered feasible if at least 12 out of 15 subjects are able to receive at least 2 weeks of tazemetostat, generate the CAR T cell product and receive CAR T cell therapy.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of DLBCL, FL, or MCL
* Eligible to receive standard of care CAR T cells
* Have received at least 1 prior therapies

Exclusion Criteria:

* Active viral infection with HIV or hepatitis type B or C
* Active, uncontrolled systemic fungal, bacterial or viral infection
* Active treatment for another cancer
* Pregnant or breastfeeding
* Unable to take oral medication
* Certain significant past medical history, such recent stroke, pulmonary embolism, myocardial infarction, congestive heart failure, uncontrolled hypertension, or certain arrhythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-10-04 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants who experience adverse events classified per CTCAEv5 | From start of treatment until 30 days after the last dose of tazemetostat, for a maximum of approximately 13 months
  Adverse reactions will be graded as per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.

SECONDARY OUTCOMES:
Number of patients who experience cytokine release syndrome (CRS) by ASTCT Consensus Grading system during therapy | From start of treatment until Day 21 days following CAR T cell infusion
  Patients will undergo screening for CRS per American Society for Transplantation and Cellular Therapy (ASTCT) guidelines
Number of patients who experience immune effector cell neurotoxicity syndrome (ICANS) by ASTCT Consensus Grading system during therapy | From start of treatment until Day 21 days following CAR T cell infusion
  Patients will undergo screening for ICANS per American Society for Transplantation and Cellular Therapy (ASTCT) guidelines
Overall response rate (ORR) reported as per Lugano response criteria | From start of treatment until disease progression or death, for a maximum of approximately 6 years
  Overall response rate will be reported as the number of participants who achieve a complete or partial response per the Lugano response criteria
Mean Progression-Free Survival (PFS) | From start of treatment until disease progression or death, for a maximum of approximately 6 years
  PFS is defined as the duration of time from start of treatment to time of documentation of progression or death from any cause.
Mean Overall Survival (OS) | From start of treatment until death, for a maximum of approximately 6 years
  OS is defined as the duration of time from start of treatment to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Yamshon, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine/NewYork-Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No